CLINICAL TRIAL: NCT00431795
Title: A Multicenter Randomized Phase II Study of Second Line Chemotherapy With Epirubicin( Farmorubicin) Versus the Pegylated Liposomal Doxorubicin in Advanced Breast Cancer Patients
Brief Title: Randomized Phase II Study of Epirubicin vs Caelyx in Pretreated Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/03.12
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: Advanced breast cancer; Pegylated liposomal doxorubicin; Epirubicin
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Epirubicin

ARMS (2):
- 1 (Experimental): Epi
  Interventions: Drug: Epirubicin
- 2 (Experimental): Cael
  Interventions: Drug: Pegylated liposomal doxorubicin (Caelyx)

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin (Caelyx) — Pegylated liposomal Doxorubicin (Caelyx) at the dose of 50mg/m^2 IV every 4 weeks for 6 consecutive cycles
  Other Names: Caelyx
  Arms: 2
Drug: Epirubicin — Epirubicin (Farmorubicin) at the dose of 90mg/m^2 IV every 3 weeks for 6 consecutive cycles
  Other Names: Farmorubicine
  Arms: 1

SUMMARY:
DOXORUBICIN is recognized as one of the most active drugs for breast cancer, but its clinical utility is limited because of a cumulative dose-dependent cardiac myopathy that can lead to potentially fatal congestive heart failure. Caelyx (pegylated liposomal doxorubicin) was designed to reduce the cardiotoxicity of doxorubicin while preserving its antitumor efficacy

DETAILED DESCRIPTION:
To compare the efficacy of pegylated liposomal doxorubicin versus epirubicin as second line chemotherapy in patient with advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate bone marrow function (Absolute neutrophil count >1000/mm^3, Platelet count>100000/mm^3, Hemoglobin>9gr/mm^3)
* Histologically- or cytologically- confirmed breast adenocarcinoma
* No prior anthracycline-based chemotherapy as treatment of advanced breast cancer
* No prior chemotherapy with ≥ 300mg/m2 doxorubicin or ≥ 540mg/m2 epirubicin as adjuvant setting
* At least 4 weeks interval since prior anticancer treatment
* Measurable disease as defined by the presence of at least one measurable lesion(except bone metastases, ascites or pleural effusions)
* Life expectancy > 3 months
* Written informed consent

Exclusion Criteria:

* Pregnancy or nursing
* Documented history of congestive heart failure (CHF), serious arrhythmia, or myocardial infarction (within 6 months)
* Other invasive malignancy except nonmelanoma skin cancer or acute infection.
* Radiation of measurable disease (except brain metastases)
* Progressive brain metastases according to clinical or radiological criteria.
* Brain metastases without prior radiation therapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Assessment of antitumor efficacy by objective tumor response rates | Objective responses confirmed by CT or MRI (on 3rd and 6th cy)

SECONDARY OUTCOMES:
Toxicity profile and tolerance between the two treatment arms | Toxicity assessment of each chemotherapy cycle
Time to progression | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki